CLINICAL TRIAL: NCT05128916
Title: Efficacy of Intralesional Platelet-rich Plasma in Treatment of Onychomycosis: a Randomized Controlled Trial
Brief Title: Efficacy of Intralesional PRP in Treatment of Onychomycosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Reem Elhaddad Ali, Assistant lecturer of Dermatology, Venereology and Andrology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OnychoPRP
Record Dates: First submitted 2021-11-11; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Platelet Rich Plasma
Keywords: PRP, platelet rich plasma, terbinafine, onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — Terbinafine

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to 3 groups. In PRP group, patients with onychomycosis will receive intralesional injections of PRP (study group 1). In PRP + terbinafine group, patients with onychomycosis will receive intralesional PRP in addition to oral terbinafine 250 mg daily (study group 2). In terbinafine group, patients with onychomycosis will receive oral terbinafine 250 mg daily (study group 3) (control group)
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of interventions (oral versus intralesional), both patient and treating investigator will not be blinded, but the assessment of outcome will be carried out by two dermatologists who will be blinded to the treatment type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intralesional PRP (Active Comparator): Patients with onychomycosis will receive intralesional injections of PRP.
  Interventions: Biological: intralesional platelet rich plasma
- Oral terbinafine (Active Comparator): Patients with onychomycosis will receive oral terbinafine 250 mg daily
  Interventions: Drug: Oral terbinafine
- Intralesional PRP + Oral terbinafine (Active Comparator): Patients with onychomycosis will receive intralesional PRP in addition to oral terbinafine 250 mg daily.
  Interventions: Biological: intralesional platelet rich plasma; Drug: Oral terbinafine

INTERVENTIONS:
Biological: intralesional platelet rich plasma — Three to fifteen milliliters of blood will be drawn from each patient then evacuated after detachment of syringe needle into 15 ml conical tube containing 3.8% sodium citrate solution. Blood will be centrifuged at 300 G-force (~ 1500 RPM) for 10 minutes. This will allow the blood to separate into 3 layers: Upper platelet-poor plasma, middle platelet-rich plasma, and lower RBCs layers. The supernatant (upper third) will be removed and the middle third (PRP) will be aspirated and used for intralesional injection of affected nails.
  Other Names: PRP
  Arms: Intralesional PRP; Intralesional PRP + Oral terbinafine
Drug: Oral terbinafine — Patients in (PRP + terbinafine) and (terbinafine) groups will receive oral 250 mg terbinafine tablets taken immediately after a fatty meal, daily for a total of 3 months
  Other Names: Terbinafine
  Arms: Intralesional PRP + Oral terbinafine; Oral terbinafine

SUMMARY:
This study aims to investigate efficacy of intralesional PRP in treatment of finer nail onychomycosis.

DETAILED DESCRIPTION:
Onychomycosis is a challenging medical condition with limited response to oral antifungal drugs. Recent study demonstrated that platelet rich plasma (PRP) have immuno-enhancing and antimicrobial properties. It had been shown that platelet microbicidal proteins released after platelet activation demonstrate potent activities against many gram-negative, gram-positive, and fungal pathogens in vitro and in vivo studies.

In addition, white blood cell concentration in PRP was reported to be two to fourfold their normal level in whole blood. Neutrophils release myeloperoxidase which has a defensive action against fungi and bacteria, while lymphocytes and monocytes both are immunogenic cells (Badade et al., 2016). Recently, PRP was successfully used in the treatment of multiple recalcitrant plane warts (Abu El-Hamd et al., 2021), Also, PRP proved its efficacy in inhibiting periodontal pathogens such as P. gingivalis and A. actinomycetemcomitans (Badade et al., 2016). In addition, relevance of platelets for antifungal defenses might be suggested by the fact that thrombocytopenia represents a highly significant risk factor for fungal infections in post-transplant liver patients (Chang et al., 2000).

This study compares between intralesional RPR versus oral antifungal versus intralesional PRP + oral antifungal in the treatment of finger nail onychmycosis.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be adult patients (> 18 years) with onychomycosis confirmed by dermoscopy, direct KOH microscopic examination and positive culture..

Exclusion Criteria:

* Patients with one or more with the following criteria will be excluded.

  1. Pregnant and lactating women.
  2. Patients received topical and/or systemic antifungal therapy during the previous 3 months.
  3. Patients with impaired liver or renal functions.
  4. Patients with anemia (hemoglobin level <10mg/dl), thrombocytopenia (platelet count < 100,000 /µL), coagulopathies or patients on anticoagulant therapy as aspirin and patients with iron deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Onychomycosis severity index | 3 months
  It is a quantitative score used to define the severity of onychomycosis. Briefly, OSI score is obtained by multiplying a score for the area of involvement (range, 0-5) by a score for the disease proximity to the matrix (range, 1-5). Ten points are added for the presence of a longitudinal streak or a patch (dermatophytoma) or greater than 2 mm of subungual hyperkeratosis. Mild onychomycosis corresponds to a score of 1- 5; moderate onychomycosis corresponds to a score of 6- 15, and severe onychomycosis corresponds to a score of 16- 35(Carney et al., 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Ramadan Saleh, MD, Study Director — Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No